CLINICAL TRIAL: NCT00729118
Title: Vorinostat (SAHA) and Lenalidomide After Autologous Transplant for Patients With Multiple Myeloma
Brief Title: Vorinostat and Lenalidomide After Autologous Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Yvonne Efebera, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08001; NCI-2011-03140 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Lenalidomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide + Vorinostat (Experimental): Maintenance post autologous transplant
  Interventions: Drug: lenalidomide; Drug: vorinostat

INTERVENTIONS:
Drug: lenalidomide — combined with Vorinostat (SAHA) days 1-21 of a 28-day cycle until progression or clinically significant toxicity.
  Other Names: Revlimid; CC-5013
Drug: vorinostat — Vorinostat (SAHA) will be administered orally beginning at dose level 1 starting day +90 ±6 days after HSCT for days 1 and 15-21 of a 28-day cycle combined with lenalidomide days 1-21 of a 28-day cycle until progression or clinically significant toxicity.
  Other Names: SAHA; Suberoylanilide hydroxamic acid

SUMMARY:
RATIONALE: Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Giving vorinostat together with lenalidomide may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat when given together with lenalidomide after autologous stem cell transplant in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the dose-limiting toxicities and safety of vorinostat and lenalidomide after autologous peripheral blood stem cell transplantation in patients with multiple myeloma.
* To evaluate the overall response rate to the combination of Vorinostat (SAHA) and lenalidomide.

Secondary

* To evaluate the effect of this treatment regimen on natural killer cell activity and regulatory T cells in the post-transplant period.
* To determine preliminary clinical activity of this treatment regimen by assessing overall survival and progression-free survival of these patients.
* To obtain pilot data regarding an association between this treatment regimen and patient quality of life and circulating inflammatory cytokines.

OUTLINE: This is a dose-escalation study of vorinostat.

Patients receive oral vorinostat alone once daily on days 1-21 in course 1. For the second and subsequent courses, patients receive oral vorinostat in combination with oral lenalidomide once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for correlative laboratory studies. Studies include functional immune assays (T-cell and natural killer cell activity and regulatory T-cell recovery) by fluorescence activated cell sorting (FACS) or ELISPOT; analysis of inflammatory markers (cytokines and catecholamines); and analysis of global H3 and H4 acetylation by immunohistochemistry.

Quality of life is assessed periodically using the Brief Pain Inventory (Short Form), The Center for Epidemiologic Studies Depression Scale (CES-D-10), a 9-item Brief Fatigue Inventory, and the FACT-G questionnaires.

After completion of study treatment, patients are followed for at least 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma
* Has undergone melphalan-conditioned autologous peripheral blood stem cell transplant myeloma.

PATIENT CHARACTERISTICS:

* ECOG/WHO performance status 0-2
* ANC ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 2 times ULN
* Serum creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 90 days after completion of study treatment
* No blood, sperm, or ova donation during and for ≥ 4 weeks after completion of study treatment
* Able to obtain commercially available lenalidomide via Celegene's RevAssist® program

  * Registered in the RevAssist® program
  * Willing and able to comply with the requirements of RevAssist®
* Able to swallow capsules
* No severe or uncontrolled systemic illness
* No "currently active" second malignancy, other than nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Patients are not considered to have a "currently active" malignancy if they completed therapy for the malignancy, are disease free from the malignancy for > 5 years, and are considered by their physician to be at < 30% risk of relapse
* No congenital long QT syndrome
* No drug or alcohol abuse within the past 12 months
* No history of allergic reactions (including erythema nodosum) attributed to compounds of similar chemical or biologic composition to lenalidomide, thalidomide, or vorinostat
* No other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the study results

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior class Ia, Ib, or Ic antiarrhythmic medication
* No prior HDAC inhibitor-like compounds (e.g., valproic acid) as anticancer therapy
* More than 30 days since prior HDAC inhibitor-like compounds for other indications (e.g., valproic acid for epilepsy)
* No prior gastrointestinal surgery or other procedure that may, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs
* No concurrent corticosteroids other than for physiologic maintenance treatment
* No concurrent radiotherapy, unless for local control of bone pain

  * Irradiated area should be as small as possible
  * Lesions within the irradiated field cannot be used for response assessment
* No concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and anticancer activity of the study drugs
* No other concurrent anticancer therapy, including chemotherapy or biologic therapy
* No other concurrent HDAC inhibitors (e.g., valproic acid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09-26 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Safety of patients receiving SAHA and lenalidomide following autologous PBSCT | up to 3 years
  Patients will be assessed for Adverse events using the NCI CTCAE version 4.0 criteria

SECONDARY OUTCOMES:
Duration of response | up to 3 years
  The time from progression to death
Time to progression (TTP) | up to 3 years
  Patients will be assessed for TTP from the start of treatment until the date of progression.
Progression-free survival (PFS) | up to 3 years
  PFS is the time from the first dose a patient receives until disease progression or death at trial closure.
Time to response | up to 3 years
  From the first dose of study therapy until measurement criteria are first met progressive response (PR), complete response (CR) or stable disease (SD). The patients best response is recorded.
Duration of overall response | up to 3 years
  The duration computed for subjects whose best response is either PR or CR or SD and is measured when first met for complete or partial response(whichever comes first) until first date of progressive disease or death
Overall survival | up to 3 years
  The survival time defined as the time from start of treatment to the date of death.
Response rate | up to 3 years
  Tumor response defined as the total number of patients whose best response is PR or CR or SD, divided by the number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne C. Efebera, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sborov DW, Benson DM, Williams N, Huang Y, Bowers MA, Humphries K, Efebera Y, Devine S, Hofmeister CC. Lenalidomide and vorinostat maintenance after autologous transplant in multiple myeloma. Br J Haematol. 2015 Oct;171(1):74-83. doi: 10.1111/bjh.13527. Epub 2015 Jun 8. PMID 26058589
- See also: Jamesline — http://cancer.osu.edu